CLINICAL TRIAL: NCT07294807
Title: Effectiveness, Safety, and Cost-effectiveness of Salt Substitution in High-risk Pregnant Women for the Prevention of Hypertensive Disorders of Pregnancy
Brief Title: Pregnancy Salt Substitution Trial for Hypertensive Disorders of Pregnancy Prevention (PREG-Salt)
Acronym: PREG-Salt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XMHEJH-WU
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Hypertensive Disorders of Pregnancy
Keywords: Sodium reduction; Pregnancy disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium-Enriched Salt substitutes (Experimental): Participants will use a potassium-enriched salt substitute in place of usual salt for home-prepared meals. The study salt substitute consists of 25% potassium chloride and 75% sodium chloride.
  Interventions: Other: Potassium-enriched salt substitute
- Usual salt (Placebo Comparator): Participants will continue to use usual salt (≥99% sodium chloride) in the preparation of home meals.
  Interventions: Other: Usual salt

INTERVENTIONS:
Other: Potassium-enriched salt substitute — replace usual salt with potassium-enriched salt containing 25% potassium chloride
  Arms: Potassium-Enriched Salt substitutes
Other: Usual salt — Usual salt (NaCl >99%)
  Arms: Usual salt

SUMMARY:
The PREG-Salt study is to evaluate the effect, safety and cost-effectiveness of low-sodium salt in reducing blood pressure and preventing hypertensive disorders in pregnant women at high risk in China. The study will recruit about 3,200 participants from approximately 100 hospitals across multiple provinces in China. Eligible pregnant women (≤16 weeks of gestation) will be randomly assigned in a 1:1 ratio to the following 2 groups:

1. Salt subsittute(intervention);
2. Usual salt (control) .

The intervention will last until delivery. The study employs an adaptive two-phase design. An interim analysis after the first phase (n=400) will inform whether the trial continues into the second phase and if any adjustments to the sample size are needed. The primary outcomes are:

Phase 1: The mean systolic blood pressure across antenatal visits (excluding the last week before delivery).

Phase 2: New-onset hypertensive disorders of pregnancy and related adverse events from randomization to delivery.

DETAILED DESCRIPTION:
The PREG-Salt study is to evaluate the effect, safety and cost-effectiveness of low-sodium salt in reducing blood pressure and preventing hypertensive disorders in pregnant women at high risk in China. Specifically, the study aims include:

1. to evaluate whether salt substitute significantly reduces mean blood pressure, while observing adherence and safety, in a high-risk population for hypertensive disorders of pregnancy.
2. to further evaluate whether salt substitute significantly reduces the incidence of hypertensive disorders of pregnancy, while assessing its safety and cost-effectiveness.

The study is a two-phase, multicenter, randomized, double-blind, parallel-group controlled study. High-risk pregnant women at ≤16 weeks of gestation will be enrolled and randomly assigned in a 1:1 ratio to either the salt substitute(intervention) group or the usual salt (control) group. The study salt will be provided free of charge until delivery. Follow-up will be conducted through all antenatal visits and delivery to collect blood pressure data and information on the incidence of hypertensive disorders of pregnancy (including gestational hypertension, preeclampsia, eclampsia, death, stillbirth, preterm birth, etc.). The study employs an adaptive design. An interim analysis will be conducted after the completion of the first phase. Based on pre-specified efficacy and safety criteria, a decision will be made regarding the continuation of the study and potential adjustments to the subsequent sample size and randomization ratio.

The study will recruit about 3,200 participants(400 participants in the first phase) from approximately 100 hospitals (with an annual delivery volume of >1,000) at the county level or above, across multiple provinces in China.

Inclusion Criteria:

1. Singleton pregnancy with a viable fetus at ≤16 weeks of gestation.
2. Meets at least one of the following criteria (enrolled sequentially):

   1. Systolic Blood Pressure (SBP) ≥130 mmHg and <160 mmHg at enrollment, OR current monotherapy with antihypertensive medications such as labetalol or nifedipine (priority enrollment).
   2. At least one of the following 4 items: advanced maternal age (≥35 years), pre-pregnancy obesity (BMI ≥28 kg/m²), history of preeclampsia, or pre-existing type 1 or type 2 diabetes.
   3. At least two of the following 5 items: history of adverse pregnancy outcome (e.g., fetal death, placental abruption, fetal growth restriction), personal history of gestational hypertension or family history of preeclampsia (mother or sister), history of gestational diabetes, obstructive sleep apnea, or pre-pregnancy overweight (BMI 24-28 kg/m²).
3. Routinely eats at least two meals per day at home (including meals brought from home).
4. Able to attend regular antenatal check-ups and is expected to complete the study follow-up.
5. Provides written informed consent.

Exclusion Criteria:

1. SBP ≥160 mmHg or Diastolic Blood Pressure (DBP) ≥110 mmHg at enrollment.
2. Conditions or history associated with high uterine tension (e.g., polyhydramnios, macrosomia, hydatidiform mole); autoimmune diseases (e.g., systemic lupus erythematosus, antiphospholipid syndrome).
3. History of chronic kidney disease, OR any antenatal check-up with a confirmed estimated Glomerular Filtration Rate (eGFR) <70 ml/min/1.73m², OR dipstick urine protein ≥2+.
4. A confirmed diagnosis of hyperkalemia.
5. History of hypotension or syncope.
6. A household member who shares meals has a confirmed diagnosis of chronic kidney disease or hyperkalemia.

Outcome Measures:

Primary outcomes:

Phase 1: Mean change in systolic blood pressure. Phase 2: New-onset Hypertensive Disorders of Pregnancy and Related Maternal Adverse Events

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy with a viable fetus at ≤16 weeks of gestation.
2. Meets at least one of the following criteria (enrolled sequentially):

   1. Systolic Blood Pressure (SBP) ≥130 mmHg and <160 mmHg at enrollment, OR current monotherapy with antihypertensive medications such as labetalol or nifedipine (priority enrollment).
   2. At least one of the following 4 items: advanced maternal age (≥35 years), pre-pregnancy obesity (BMI ≥28 kg/m²), history of preeclampsia, or pre-existing type 1 or type 2 diabetes.
   3. At least two of the following 5 items: history of adverse pregnancy outcome (e.g., fetal death, placental abruption, fetal growth restriction), personal history of gestational hypertension or family history of preeclampsia (mother or sister), history of gestational diabetes, obstructive sleep apnea, or pre-pregnancy overweight (BMI 24-28 kg/m²).
3. Routinely eats at least two meals per day at home (including meals brought from home).
4. Able to attend regular antenatal check-ups and is expected to complete the study follow-up.
5. Provides written informed consent. -

Exclusion Criteria:

1. SBP ≥160 mmHg or Diastolic Blood Pressure (DBP) ≥110 mmHg at enrollment.
2. Conditions or history associated with high uterine tension (e.g., polyhydramnios, macrosomia, hydatidiform mole); autoimmune diseases (e.g., systemic lupus erythematosus, antiphospholipid syndrome).
3. History of chronic kidney disease, OR any antenatal check-up with a confirmed estimated Glomerular Filtration Rate (eGFR) <70 ml/min/1.73m², OR dipstick urine protein ≥2+.
4. Diagnosed hyperkalemia.
5. History of hypotension or syncope.
6. A household member who shares meals has a confirmed diagnosis of chronic kidney disease or hyperkalemia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-25 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | from baseline to 36-37 weeks of gestation
  Mean change in systolic blood pressure across antenatal visits (excluding the week before delivery) during the follow-up period.
Incidence of new-onset hypertensive disorders of pregnancy and related maternal adverse events | from randomization to delivery
  A prespecified hierarchical composite endpoint including the first occurrence of any of the following events from randomization to delivery: 1）Maternal death or pregnancy loss; 2）New-onset preeclampsia, eclampsia, or placental abruption; 3）New-onset gestational hypertension or clinically meaningful elevation in blood pressure meeting diagnostic criteria.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure | from baseline to 36-37 weeks of gestation
  Mean change in diastolic blood pressure across antenatal visits (excluding the week before delivery) during the follow-up period.
Incidence of new-onset hypertensive disorders of pregnancy | from randomization to delivery
  hypertensive disorders of pregnancy is defined as a baseline blood pressure <140/90 mmHg without antihypertensive medication, followed by any two consecutive measurements of systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg during follow-up, or the initiation of antihypertensive medication under a physician's guidance.
Incidence of clinically meaningful increase in blood pressure | from randomization to delivery
  Clinically meaningful increase in blood pressure is defined as an average systolic blood pressure increase of >10 mmHg from baseline, measured at any two consecutive follow-up visits, in participants with a baseline blood pressure ≥140/90 mmHg or those receiving antihypertensive therapy.
Incidence of preeclampsia or eclampsia | from randomization to delivery
  Preeclampsia is defined as the presence of gestational hypertension or chronic hypertension in pregnancy, accompanied by any one of the following: a 24-hour urinary protein excretion ≥0.3 g; a urinary albumin-to-creatinine ratio ≥0.3, a random urine protein ≥1+(for patients with chronic hypertension and pre-existing baseline proteinuria, in the absence of organ dysfunction, the diagnosis of superimposed preeclampsia requires a doubling of the proteinuria level (either 24-hour urinary protein or urinary microalbumin-to-creatinine ratio) from the baseline); no proteinuria but accompanied by any of the following organ or system involvement(cardiac, pulmonary, hepatic, renal, hematologic, digestive, or nervous system, or evidence of placental-fetal involvement).
  Eclampsia is defined as the occurrence of new-onset, tonic-clonic seizures in a woman with preeclampsia, which cannot be attributed to other explainable causes.
Incidence of maternal death | from randomization to delivery
  death during the study period resulting from any pregnancy-related or aggravated condition, excluding deaths from accidental or incidental causes, determined based on death records in hospital medical records or death certificates.
Incidence of pregnancy loss | from randomization to delivery
  Pregnancy loss is defined as any of the following situations: spontaneous abortion, fetal death, stillbirth, medically Induced abortion or termination of pregnancy, neonatal death
Incidence of Placental abruption | from randomization to delivery
  Placental abruption is defined as the partial or complete separation of the placenta from the uterine wall before the delivery of the fetus. It is characterized by sudden onset abdominal pain, vaginal bleeding, uterine tenderness, and/or fetal distress. The diagnosis is confirmed by the discharge diagnosis or operative records.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | from randomization to delivery
  all causes adverse events
Incidence of all-cause maternal mortality | from randomization to delivery
  All-cause mortality, regardless of its association with pregnancy or childbirth.
Incidence of hyperkalemia | from randomization to delivery
  Hyperkalemia is defined as a follow-up serum potassium level >5.5 mmol/L accompanied by pathological ECG changes, persistent serum potassium >5.5 mmol/L, or hyperkalemia diagnosed by a clinician during the study period.
Incidence of sudden cardiac death | from randomization to delivery
  Sudden cardiac death is defined as unexpected natural death due to cardiac causes, occurring within one hour of symptom onset in a person with or without known pre-existing heart disease
Incidence of hyponatremia | from randomization to delivery
  Hyponatremia is defined as a follow-up serum sodium level <135 mmol/L, or hyponatremia diagnosed by a clinician during the study period.
Incidence of renal impairment | from randomization to delivery
  Renal impairment is defined as urinary protein quantification >2.0 g/24 h, or UACR ≥2000 mg/g in any follow-up or during the study period; or serum creatinine level >106 μmol/L.
Incidence of hypotension | from randomization to delivery
  Hypotension is defined as at least two blood pressure readings <90/60 mm Hg during follow-up, or symptomatic hypotension diagnosed by a physician during treatment.
Incremental Cost-Effectiveness Ratio (ICER) | from randomization to delivery
  Incremental Cost-Effectiveness Ratio (ICER) is defined as (Intervention Group Cost - Control Group Cost) / (Intervention Group Effectiveness - Control Group Effectiveness).
Incidence of preterm birth | At delivery
  preterm birth is defined as the delivery of a live-born infant before 37 completed weeks of gestation, including both medically indicated and spontaneous preterm births, confirmed by hospital medical records, surgical notes, or discharge diagnoses.
Gestational age at delivery | At delivery
  Gestational age at delivery
The neonatal birth weight | At delivery
  Birth weight of the newborn
Incidence of neonatal adverse outcomes | delivery
  Neonatal adverse outcomes include neonatal intensive care unit (NICU) admission, small for gestational age (SGA), and severe neonatal complications.
Mean change in Insomnia Severity Index (ISI) score | From baseline to 36-37 weeks of gestation
  Insomnia Severity Index (ISI) score is a patient-reported outcome assessing insomnia severity, with higher scores indicating more severe insomnia.
Mean change in spot urinary potassium | From baseline to 30-32 weeks of gestation
  Spot urinary potassium concentration, used as a proxy indicator of dietary potassium intake.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Principal Investigator — Peking University; Yangfeng Wu, Principal Investigator — Peking University
Locations (107):
- China (107):
  - Chongqing Bishan District Maternal and Child Health Care Hospital, Bishan, Chongqing Municipality
  - Chongqing Fuling District Maternal and Child Health Care Hospital, Fuling, Chongqing Municipality
  - Chongqing Qijiang District People's Hospital, Gunan, Chongqing Municipality
  - Chongqing Hechuan District Maternal and Child Health Care Hospital, Hechuan, Chongqing Municipality
  - Chongqing Jiangjin District Maternal and Child Health Care Hospital, Jiangjin, Chongqing Municipality
  - Chongqing Qianjiang District Maternal and Child Health Care Hospital, Qianjiang, Chongqing Municipality
  - The First Affiliated Hospital of Army Medical University (Xinan Hospital), Shapingba, Chongqing Municipality
  - The Second Affiliated Hospital of Army Medical University (Xinqiao Hospital), Shapingba, Chongqing Municipality
  - University Town Hospital of Chongqing Medical University, Shapingba, Chongqing Municipality
  - Chongqing Wulong District Maternal and Child Health Care Hospital, Wulong, Chongqing Municipality
  - Chongqing Wushan County People's Hospital, Wushan, Chongqing Municipality
  - Chongqing Yongchuan District Maternal and Child Health Care Hospital, Yongchuan, Chongqing Municipality
  - Chongqing Maternal and Child Health Care Hospital, Yubei, Chongqing Municipality
  - Chongqing Yubei District Maternal and Child Health Care Hospital, Yubei, Chongqing Municipality
  - Chongqing Yunyang County People's Hospital, Yunyang, Chongqing Municipality
  - Army Specialty Medical Center (Daping Hospital), Yuzhong, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Baoding Maternal and Child Health Hospital, Baoding, Hebei
  - Yixian Maternal and Child Health Hospital, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Cangzhou Maternal and Child Health Hospital, Cangzhou, Hebei
  - Huanghua People's Hospital, Cangzhou, Hebei
  - Gucheng County Hospital, Hengshui, Hebei
  - Hengshui Fourth Hospital, Hengshui, Hebei
  - Hengshui Maternal and Child Health Care Hospital, Hengshui, Hebei
  - China Petroleum Central Hospital (Hebei), Langfang, Hebei
  - Hebei Yanda Hospital, Langfang, Hebei
  - Langfang People's Hospital, Langfang, Hebei
  - Qinhuangdao Changli County Maternal and Child Health Hospital, Qinhuangdao, Hebei
  - Qinhuangdao Maternal and Child Health Hospital, Qinhuangdao, Hebei
  - Qinhuangdao Qinglong County People's Hospital, Qinhuangdao, Hebei
  - Shijiazhuang Maternity & Child Healthcare Hospital, Shijiazhuang, Hebei
  - Xinle City Hospital, Shijiazhuang, Hebei
  - Linxi County People's Hospital, Xingtai, Hebei
  - Weixian County People's Hospital, Xingtai, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Guyuan Maternal and Child Health Care Hospital, Guyuan, Ningxia
  - Guyuan People's Hospital, Guyuan, Ningxia
  - Lingwu People's Hospital, Lingwu, Ningxia
  - Pingluo County People's Hospital, Pingluo Chengguanzhen, Ningxia
  - Shizuishan First People's Hospital, Shizuishan, Ningxia
  - Wuzhong People's Hospital, Wuzhong, Ningxia
  - Ningxia Hui Autonomous Region Hospital of Traditional Chinese Medicine, Xixia, Ningxia
  - Ningxia Hui Autonomous Region People's Hospital, Yinchuan, Ningxia
  - Peking University First Hospital Ningxia Women and Children's Hospital, Yinchuan, Ningxia
  - Yinchuan First People's Hospital, Yinchuan, Ningxia
  - Yinchuan Maternal and Child Health Care Hospital, Yinchuan, Ningxia
  - Tongxin County People's Hospital, Yuhai, Ningxia
  - Zhongning County People's Hospital, Zhongwei, Ningxia
  - Zhongwei People's Hospital, Zhongwei, Ningxia
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University (Dezhou Hospital), Dezhou, Shandong
  - Dongying Second People's Hospital, Dongying, Shandong
  - Dong'e County People's Hospital, Dong’e, Shandong
  - Feicheng People's Hospital, Feicheng, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Jinan Maternal and Child Health Care Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Maternal and Child Health Care Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital), Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - The Second Jinan Maternal and Child Health Care Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - The Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Laizhou Maternal and Child Health Hospital, Laizhou, Shandong
  - Lanling County People's Hospital, Lanling, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Chengyang District People's Hospital, Qingdao, Shandong
  - Qingdao Women and Children's Hospital (Peking University People's Hospital Qingdao Branch), Qingdao, Shandong
  - Rizhao People's Hospital, Rizhao, Shandong
  - Taian Central Hospital, Taian, Shandong
  - Weifang Maternal and Child Health Hospital, Weifang, Shandong
  - Weihai Maternal and Child Health Hospital, Weihai, Shandong
  - Yantai Yeda Hospital, Yantai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Rongcheng Maternal and Child Health Hospital, Yatou, Shandong
  - Zaozhuang Maternal and Child Health Hospital, Zaozhuang, Shandong
  - Huantai County Maternal and Child Health Hospital, Zibo, Shandong
  - Zibo Maternal and Child Health Hospital, Zibo, Shandong
  - Zoucheng People's Hospital, Zoucheng, Shandong
  - Zouping People's Hospital, Zouping, Shandong
  - Xinjiang Military Region General Hospital, Ürümqi, Xingjiang
  - The First People's Hospital of Aksu Prefecture, Aksu, Xinjiang
  - Altay Prefecture People's Hospital, Altay, Xinjiang
  - Kizilsu Kirgiz Autonomous Prefecture People's Hospital, Artux, Xinjiang
  - Bortala Mongolian Autonomous Prefecture People's Hospital, Bole, Xinjiang
  - Changji Hui Autonomous Prefecture People's Hospital, Changji, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University (Changji Branch), Changji, Xinjiang
  - Hami Central Hospital, Hami, Xinjiang
  - Hotan Prefecture People's Hospital, Hotan, Xinjiang
  - Karamay Central Hospital, Karamay, Xinjiang
  - The First People's Hospital of Kashi, Kashgar, Xinjiang
  - The Second People's Hospital of Kashi Prefecture, Kashgar, Xinjiang
  - Bayingolin Mongolian Autonomous Prefecture People's Hospital, Korla, Xinjiang
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - Turpan Gaochang District People's Hospital, Turpan, Xinjiang
  - Turpan People's Hospital, Turpan, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Urumqi First People's Hospital (Railway Bureau Campus), Ürümqi, Xinjiang
  - Urumqi Maternal and Child Health Care Hospital (Urumqi You'ai Hospital), Ürümqi, Xinjiang
  - Yili Prefecture Friendship Hospital, Yining, Xinjiang
  - Chongqing Wanzhou District Maternal and Child Health Care Hospital, Wanzhou

IPD SHARING:
Plan to Share IPD: Yes